CLINICAL TRIAL: NCT02207842
Title: The Determination of the Effect of Volatile Anesthetics on Leukocyte Function ex Vivo
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, staff anesthesiologist, Boston Children's Hospital
Other Study IDs: P00012751
Record Dates: First submitted 2014-07-30; First posted 2014-08-04 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Leukocyte Function; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Volatile anesthesia exposure
- No volatile anesthesia exposure

SUMMARY:
One of the most common side effects of a surgical procedure is infection. In order to lower the number of infections that occur after surgery, it is important for physicians to know how medications used during surgery affect the way the body fights infection. Often, when anesthesiologists are helping people go to sleep before surgery they give people medications known as "volatile anesthetics". Volatile anesthetics are medications that can change from a liquid or solid to a gas very easily. Some studies suggest that these types of medications may change the way white blood cells work in the body. Changing the way white blood cells work could possibly increase the person's risk of infection after their surgery or weaken their body's ability to fight infections. The goal of this research study is to learn about how volatile anesthesia medications change the way white blood cells work in people having anesthesia for cardiac procedures. To do this, investigators will examine the function of while blood cells in the laboratory based setting.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* greater than or equal to 12 months of age
* scheduled for a cardiac catheterization, cardiac surgery, or cardiac MRI

Exclusion Criteria:

* known underlying hematological disorder
* known oncological disorder
* patients who do not require preoperative laboratory testing

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients greater than or equal to 12 months of age, who present for a cardiac catheterization, cardiac surgery, or cardiac MRI at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Leukocyte function under anesthesia | up to 12 months
  The study will evaluate ex vivo leukocyte function by testing leukocyte activation, TNF-a production, and phagocytic function in the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Yuki, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States